CLINICAL TRIAL: NCT03534492
Title: Impact of the Combination of Durvalumab (MEDI4736) Plus Olaparib (AZD2281) Administered Prior to Surgery in the Molecular Profile of Resectable Urothelial Bladder Cancer.
Brief Title: Durvalumab Plus Olaparib Administered Prior to Surgery of Resectable Urothelial Bladder Cancer (NEODURVARIB)
Acronym: NEODURVARIB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Oncology Genito-Urinary Group (Other)
Collaborators: AstraZeneca (Industry); Sistemas Genómicos (Unknown); Apices Soluciones S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOGUG-2017-A-IEC(VEJ)-2; 2017-002765-22 (EudraCT Number)
Record Dates: First submitted 2018-05-11; First posted 2018-05-23 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Bladder Cancer
Keywords: urothelial; bladder cancer; olaparib; durvalumab
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — durvalumab; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab plus Olaparib (Experimental): Durvalumab 1500 mg every 4 weeks for up to a maximum of 2 months (up to 2 doses/cycles) plus Olaparib 300 mg b.i.d. up to 56 days (2 cycles of 28 days each cycle).
  Interventions: Drug: Durvalumab; Drug: Olaparib

INTERVENTIONS:
Drug: Durvalumab — Infusion
Drug: Olaparib — P.O.

SUMMARY:
The standard of care for muscle-invasive bladder cancer (MIBC) is radical cystectomy, which is rarely curative. Platinum-based neoadjuvant chemotherapy is associated with an improvement in Overall Survival (OS), but only a few patients can benefit from this approach. Therefore, new neoadjuvant treatments are required for muscle- invasive bladder cancer. In this study it will be explored the activity of durvalumab plus olaparib in advanced Transitional Cell Carcinoma of the Bladder and therefore may have beneficial outcomes in the neoadjuvant setting. Adverse events associated with durvalumab and olaparib is one of the potential risks in this study. Participation in this trial, in which 6-8 weeks of preoperative treatment will be administered, is not expected to result in delays of surgery for participants. It is not foreseen that treatment with durvalumab and olaparib has a relevant impact on operability or increases the risks associated with surgery

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the subject prior to performing any protocol related procedures, including screening evaluations
2. Age ≥18 years at time of study entry
3. Subjects with histological confirmation of T2-T4a urothelial bladder by transurethral resection
4. Patients aimed for cystectomy without neoadjuvant chemotherapy
5. Tumor tissue (archival or recent acquisition) from diagnostic Transurethral Resection (TUR) must be available (block or 5 - 15 unstained slides of formalin fixed paraffin embedded (FFPE) tissue) for correlative studies.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 Exclusion Criteria.
7. Life expectancy of > 16 weeks
8. Body weight > 30kg
9. Normal organ and bone marrow function prior to administration of study treatment as defined below:

   * Haemoglobin > 10.0 g/dL with no blood transfusion in the past 28 days
   * Absolute neutrophil count (ANC) 1.5 x (> 1500 per mm3)
   * Platelet count ≥ 100 x 109/L (>100,000 per mm3)
   * Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN).
   * Aspartate aminotransferase (AST)/ alanine aminotransferase (ALT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤ 5x ULN
   * Serum creatinine Clearance > 51 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance.
10. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal subjects within 28 days of study treatment and confirmed prior to treatment on day 1.
11. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.
12. Male patients and their partners, who are sexually active and of childbearing potential, must agree to the use of two highly effective forms of contraception in combination, throughout the period of taking study treatment and for 180 days after last dose of study drug(s) to prevent pregnancy in a partner. Female patients of child bearing potential and male patients with partners of child bearing potential, who are sexually active, must agree to the use of two highly effective forms of contraception throughout period of taking study treatment and for 1 month (female patients) / 3 months (male patients) after last dose of study drug.
13. At least one lesion (measurable and/or non-measurable) that can be accurately assessed at baseline by CT/MRI and is suitable for repeated assessment.
14. Formalin fixed, paraffin embedded (FFPE) tumour sample from the primary cancer must be available for central testing. If there is not confirmation of the availability of an archived tumour sample prior to enrolment the patient is not eligible for the study

Exclusion criteria:

1. Participation in another clinical study with an investigational product during the last 4 weeks
2. Concurrent enrolment in another clinical study, unless it is an observational (non- interventional) clinical study or during the follow-up period of an interventional study
3. Prior therapy with anti-PD-1, anti-PD-L1 including durvalumab, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody (or any other antibody or drug specifically targeting T-cell co- stimulation or checkpoint pathways).
4. Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) ≤ 28 days prior to the first dose of study drug.
5. Resting electrocardiogram (ECG) with time between the start of the Q wave and the end of the T wave corrected for heart rate (QTc)> 470 msec on 2 or more time points within a 24 hour period or family history of long QT syndrome.
6. Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid.
7. Any unresolved toxicity National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Grade ≥1 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria
8. Any concurrent chemotherapy, Investigational Product (IP), biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (eg, hormone replacement therapy) is acceptable.
9. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug.
10. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP and patients must have recovered from any effects of any major surgery.
11. Previous allogenic bone marrow transplant or double umbilical cord blood transplant (dUCBT).
12. Whole blood transfusions in the last 120 days prior to entry to the study (packed red blood cells and platelet transfusions are acceptable.
13. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]).
14. Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non- malignant systemic disease or active, uncontrolled infection.
15. Past medical history of Interstitial Lung Disease (ILD), drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.
16. Subjects with uncontrolled adrenal insufficiency
17. Known drug or alcohol abuse
18. History of another primary malignancy.
19. Patients with symptomatic uncontrolled brain metastases.
20. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis (TB) testing in line with local practice), hepatitis B (known positive Hepatitis B Virus (HBV) surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Subjects with a past or resolved HBV infection (defined as the presence of hepatitis B core (HBc) antibody [anti-HBc] and absence of HBsAg) are eligible. Subjects positive for hepatitis C, HIV, or immunocompromised patients are eligible only if polymerase chain reaction is negative for Hepatitis C Virus (HCV) RNA.
21. Receipt of live attenuated vaccine within 30 days prior to the first dose of study treatment.
22. Female subjects who are pregnant or breastfeeding or male or female subjects of reproductive potential who are not willing to employ effective birth control from screening to 180 days after the last dose of study treatment.
23. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
24. Prior randomisation or treatment in a previous durvalumab and/or tremelimumab clinical study regardless of treatment arm assignment.
25. Prisoners or subjects who are involuntarily incarcerated.
26. Any previous treatment with poly ADP ribose polymerase (PARP) inhibitor, including olaparib.
27. Concomitant use of known strong CYP3A inhibitors (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks.
28. Concomitant use of known strong (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
29. Patients with myelodysplastic syndrome/acute myeloid leukaemia or with features suggestive of MyeloDysplatic Syndrome (MDS) / acute myeloid leukemia (AML).
30. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
31. Judgment by the investigator that the patient is unsuitable to participate in the study
32. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
33. Previous enrolment in the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Impact of neoadjuvant treatment with durvalumab plus olaparib in the molecular profile of resectable urothelial bladder cancer (Pathological complete response rate (pCRR)) | 24 weeks
  pCRR will be analysed based on the percentage of patients who obtained a pathological complete response. Pathologic response will be evaluated on cystectomy tumor sample

SECONDARY OUTCOMES:
Radiological response of durvalumab plus olaparib as presurgical treatment | 16 weeks
  Radiological response will be assessed according to RECIST 1.1 criteria in patients with measurable and/or non-measurable disease at baseline that can be accurately assessed at baseline by computed tomography (CT) / magnetic resonance imaging (MRI) and is suitable for repeated assessment and previous to cystectomy. Patients without a radiologic post-baseline tumour assessment will be considered not evaluable for this endpoint.
Toxicity profile of durvalumab plus olaparib as presurgical treatment in bladder cancer | 28 weeks
  Percentage of patients with each of the adverse event per grade

OTHER OUTCOMES:
Predictive and prognostic exploratory biomarkers in collected tumour tissue and plasma and their association with disease status and/or response/failure to study treatment | 24 weeks
  Summary statistics and corresponding changes (or percent changes) from baseline tabulated by time and cohort

CONTACTS AND LOCATIONS:
Overall Officials: Jesús García-Donas, MD PhD, Principal Investigator — Centro Integral Oncológico Clara Campal; Juan F Rodriguez-Moreno, MD, Principal Investigator — Centro Integral Oncológico Clara Campal
Locations (10):
- Spain (10):
  - ICO Badalona, Badalona, Barcelona
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Clinica IMQ Zorrotzaurre, Bilbao
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Ramón Y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hopsital Universitario Madrid Sanchinarro (CIOCC), Madrid
  - Hospital de Navarra, Pamplona
  - Hospital Virgen Macarena, Seville

IPD SHARING:
Plan to Share IPD: No